CLINICAL TRIAL: NCT04612036
Title: Multi-center In Vivo Kinematics for Subjects Implanted With Smith & Nephew Journey II BCS TKA, Journey II CR TKA, Or Journey II XR TKA
Brief Title: In Vivo Kinematics for Subjects With Smith & Nephew Journey II BCS TKA, Journey II CR TKA, Or Journey II XR TKA
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Other Study IDs: WIRB20203268
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplasty; Knee
Keywords: Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Journey II Bi-Cruciate Stabilized: Subjects who have received a Journey II Total Knee Arthroplasty with both the ACL and PCL resected
  Interventions: Device: Journey II Bi-Cruciate Stabilized TKA
- Journey II Cruciate Retaining: Subjects who have received a Journey II Total Knee Arthroplasty with only the ACL resected (therefore PCL retained)
  Interventions: Device: Journey II Cruciate Retaining TKA
- Journey II Bi-Cruciate Retaining: Subjects who have received a Journey II Total Knee Arthroplasty with both the ACL and PCL retained
  Interventions: Device: Journey II Bi-Cruciate Retaining TKA

INTERVENTIONS:
Device: Journey II Bi-Cruciate Stabilized TKA — Total Knee Arthroplasty System
  Groups: Journey II Bi-Cruciate Stabilized
Device: Journey II Cruciate Retaining TKA — Total Knee Arthroplasty System
  Groups: Journey II Cruciate Retaining
Device: Journey II Bi-Cruciate Retaining TKA — Total Knee Arthroplasty System
  Groups: Journey II Bi-Cruciate Retaining

SUMMARY:
The objective of this study is to determine and compare the in vivo kinematics and vibroarthrography (VAG) signals for subjects implanted with Journey II Bi-Cruciate Stabilized (BCS), CR (Cruciate Retaining), and Bi-Cruciate Retaining (XR) TKAs.

DETAILED DESCRIPTION:
The objective of this study is to determine and compare the in vivo kinematics and vibroarthrography (VAG) signals for subjects implanted with Journey II Bi-Cruciate Stabilized (BCS), CR (Cruciate Retaining), and Bi-Cruciate Retaining (XR) TKAs. The Journey II BCS Knee System was designed to resect and replicate both the PCL and ACL, the Journey II CR System retains the posterior cruciate ligament, while the Journey II XR System retains the cruciate and collateral ligaments so they remain intact.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the age range of 18 years to 85 years (both inclusive)
2. Patients who have a BMI less than 35
3. Patients who do not have previous surgery on the implanted knee that might restrict their movement
4. Patient who are at least 6 months post-operative
5. Patients who do not experience any pain or other post-operative complications
6. Patients who have a stable TKA and can perform a deep knee bend activity
7. Patients who are willing to participate in this study and are willing to sign appropriate HIPAA and informed consent forms
8. Subjects will have a Journey II, either the BCS or XR, knee system

Exclusion Criteria:

1. Pregnant, potentially pregnant, or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
2. Patients who have currently enrolled in a fluoroscopic study within the past year.
3. Patients currently involved in any personal injury litigation, medical/legal or workman's compensation claims.
4. Patients with known drug or alcohol abuse histories or psychological disorders that could affect ability to complete all aspects of the study.
5. Patients with neurological or musculoskeletal disorders that might adversely affect weight-bearing motion ability
6. Subjects who are unable to perform a deep knee bend.
7. Subjects who are unwilling to sign Informed Consent/ HIPAA documents.
8. Subjects without the required type of knee implant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Journey II Bi-Cruciate Stabilized (BCS), CR (Cruciate Retaining), and Bi-Cruciate Retaining (XR) TKAs
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael LaCour, PhD, Principal Investigator — The University of Tennessee
Locations (1):
- The University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Researchers would like to retain this study data in our secure database so as to continue to add relevant, current data to our digital collection to help us work with manufacturers in the future to create better implants that last longer and will not require revision surgery. Participants will be asked if their study data may remain a part of the University of Tennessee's Center for Musculoskeletal Research data collection for use in future studies in the IC. Identifiers are automatically removed from the database upon entry into the secure server. Data shared with sponsors is de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
Started | 25 | 25 | 10
Completed | 25 | 25 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining | Total
Number analyzed (Participants) | 25 | 25 | 10 | 60
Age, Customized [Count of Participants; unit: Participants]
  <18 | 0 | 0 | 0 | 0
  18-85 | 25 | 25 | 10 | 60
  85+ | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 5 | 40
  Male | 7 | 8 | 5 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Medial AP Translations, in mm
Description: Anterior Posterior (AP) translations, in mm, of medial femoral condyle during Deep Knee Bend Activity. Values are based on the participants range of motion throughout their DKB activity. A positive number indicated anterior sliding from full extension to maximum flexion, and a negative number indicated posterior rollback from full extension to maximum flexion.
Time Frame: At least 6 months postoperative
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
Number analyzed (Participants) | 25 | 25 | 10
millimeters | -6.9 (2.8) | -0.2 (4.3) | -4.4 (3.8)

2. Primary Outcome: Lateral AP Translations, in mm
Description: Anterior Posterior (AP) translations, in mm, of lateral femoral condyle during Deep Knee Bend Activity. Values are based on the participants range of motion throughout their DKB activity. A positive number indicated anterior sliding from full extension to maximum flexion, and a negative number indicated posterior rollback from full extension to maximum flexion.
Time Frame: At least 6 months postoperative
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
Number analyzed (Participants) | 25 | 25 | 10
millimeters | -12.5 (5.0) | -4.7 (6.2) | -9.4 (6.1)

3. Primary Outcome: Maximum Flexion, in Degrees
Description: Maximum weight-bearing flexion, in degrees, during Deep Knee Bend Activity. Maximum flexion indicated how far a participant can bend their knee during a DKB. A larger number indicates greater flexion, i.e. more bending.
Time Frame: At least 6 months postoperative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
Number analyzed (Participants) | 25 | 25 | 10
degrees | 108 (13) | 121 (6) | 105 (13)

4. Primary Outcome: Axial Rotation, in Degrees
Description: Axial Rotation, in degrees, during Deep Knee Bend Activity. Values are based on the participants range of motion throughout their squat activity. A positive number indicates external femorotibial axial rotation from full extension to maximum flexion, and a negative number indicates internal femorotibial axial rotation from full extension to maximum flexion.
Time Frame: At least 6 months postoperative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
Number analyzed (Participants) | 25 | 25 | 10
degrees | 7.1 (4.2) | 5.6 (5.7) | 6.0 (7.0)

ADVERSE EVENTS:
Time Frame: adverse events would be noted on day of data collection. therefore the adverse events would be noted immediately, i.e. 1 day.
Arm/Group | Journey II Bi-Cruciate Stabilized | Journey II Cruciate Retaining | Journey II Bi-Cruciate Retaining
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/10
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04612036/Prot_SAP_000.pdf